CLINICAL TRIAL: NCT03329625
Title: PREVENTING CONDUCT DISORDER AMONG CHILDREN IN THE CHILD WELFARE SYSTEM
Brief Title: Preventing Conduct Disorder in Child Welfare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Patricia Kohl, Ph.D., Associate Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R01HD061454 (NIH)
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Behavioral Disorder; Child Maltreatment
Keywords: Triple P; RCT; parent management training; Child welfare; child behavior problems
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pathways Triple P (Experimental): Families randomized to the Pathways Triple P received a 14 week home based intervention.
  Interventions: Behavioral: Pathways Triple P
- Services as Usual (Active Comparator): Families randomized to the services as usual condition received services as usual through the Missouri Children's Division
  Interventions: Behavioral: Services as Usual

INTERVENTIONS:
Behavioral: Pathways Triple P — Pathways Triple was developed by Matt Sanders and is a behavioral parent training intervention designed to treat child behavior problems and prevent child maltreatment.
  Arms: Pathways Triple P
Behavioral: Services as Usual — Families received family centered services and other parenting interventions as deemed appropriate by the child welfare case manager.
  Arms: Services as Usual

SUMMARY:
A mixed methods randomized control trial was conducted to test the effectiveness of Pathways Triple P with child welfare involved families compared to treatment as usual. Outcomes tested included parenting behaviors and attitudes, and child behavior problems. 144 families were recruited into the study. Data was collected at 4 time points (baseline, 4 months, 9 months, and 18 months). Over 70% were retained from baseline to 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Families with open child protective service case following allegation of child physical abuse or neglect
* parent of child between the age of 3 and 12
* Child remained in the home following investigation
* parent spoke English

Exclusion Criteria:

* parent's child could not have chronic medical condition or have a pervasive developmental delay

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2010-07-05 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Eyberg Child Behavior Inventory | 18 months
  Child Behavior Problems
PedsQL | 18 months
  Pediatric Quality of Life Scale

SECONDARY OUTCOMES:
Parenting Stress Inventory | 18 months
  Parent Stress
Parent Anger Inventory | 18 months
  Parent Anger
Parental Sense of Competence | 18 months
  Parent Sense of Competence
Alabama Parenting Questionnaire | 18 months
  Parenting Behavior Inventory
Depression Anxiety Stress Scales | 18 months
  Parental Mental Health
AUDIT | 18 months
  Alcohol Abuse in Parents
The Drug Abuse Screening Test | 18 months
  Parent Substance use
HITS IPV Screening | 18 months
  Domestic Violence history
PQL | 18 months
  Parent Report of Child Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Kohl, PhD, Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No